CLINICAL TRIAL: NCT04457401
Title: The Effect of a Probiotic on Gastrointestinal Symptoms Due to Menstruation in Healthy Adult Women: a Randomized, Double-blind, Controlled Clinical Trial
Brief Title: Probiotic and Gastrointestinal Symptoms Due to Menstruation in Healthy Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB201901746
Record Dates: First submitted 2020-06-17; First posted 2020-07-07 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Menstrual Discomfort
Keywords: Gastrointestinal function
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled parallel study in which participants receive one of the study supplements (probiotic or placebo) for an 8-week intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants, investigators, and anyone else directly involved with the study will remain blinded for its entirety.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): 1 capsule daily for 8 weeks, containing 3 x 10^9 colony forming units/capsule of a Bifidobacterium strain
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): 1 capsule daily for 8 weeks containing the same carrier material and is similar in size, shape and taste to probiotic
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — This probiotic is commercially available and contains Bifidobacterium (3 x 10^9 colony forming units/capsule) as the active ingredient and potato starch, magnesium stearate and ascorbic acid as excipients.
  Arms: Probiotic
Dietary Supplement: Placebo — The placebo contains potato starch, magnesium stearate and ascorbic acid.
  Arms: Placebo

SUMMARY:
In this double blind, parallel study, female participants who are on an oral contraceptive will consume either a probiotic or placebo supplement for approximately 8 weeks. Menstrual cramp and abdominal pain severity, as measured by the visual analog scale, will be assessed daily. A subgroup of participants will be asked to provide vaginal swab and stool samples to assess microbial communities.

DETAILED DESCRIPTION:
Participants recruited from the university community in the Southeast U.S. will participate in a randomized, double-blind, placebo-controlled interventional study for approximately 8 weeks following obtainment of informed consent. Participants will be asked to maintain their usual physical activity level as well as their usual diets with the exception of fermented foods, food containing added probiotics (e.g. yogurts with live, active cultures or supplements or probiotic supplements), or foods with added fiber supplements.

After obtaining consent, participants will be randomized to receive either the probiotic or placebo daily for 8 weeks. All study days will be ± 3 days to account for variation in each participant's menstrual cycle. The study supplements will be distributed approximately 7 days before their first menstrual event. Participants will be instructed to begin taking the study supplement 3 days after they menstruate.

At randomization, participants will be asked to start completing daily questionnaires inquiring about gastrointestinal symptoms, abdominal pain as measured by a visual analog scale, duration of abdominal pain, stool form and number, adverse events, and medications taken, including the dose and administration schedule. On the third day of their menstrual cycle (day 3/menstruation 1), they will begin consuming their study supplement (start of intervention). On the days participants experience gastrointestinal symptoms related to the menstrual cycle, they will answer an additional questionnaire asking about gastrointestinal symptoms. Approximately seven days prior to the first menstrual cycle (study day -7) and three days after each menstrual event (study day 3 and 31), participants will answer the Menstrual Symptom Questionnaire to assess symptoms leading up to and during menstruation. Seven days after each menstrual event (study days 7 and 35), participants will be administered the Perceived Stress Scale to assess stress levels over the previous month. Participants will also answer two validated weekly questionnaires inquiring about gastrointestinal symptoms and how symptoms affect quality of life each week they are in the study. Each participant will also complete a 24-hour dietary recall assessment at four points during the study (study day -7, 21, 28, and 35) in order to determine how dietary patterns fluctuate throughout the menstrual cycle. A subgroup of participants will be asked to provide six additional vaginal swab and stool samples and six additional dietary recalls.

A subgroup of 20 participants per arm will also be consented to provide ten stool samples and vaginal swabs during the study (study day -7, 1, 7, 14, 21, 28, 35, 42, 49, & 56). Participants will be provided with stool and vaginal swab collection kits. Participants will self collect both of these samples and may either collect them at home or may use a restroom in the Food Science and Human Nutrition building to self collect. Coolers will be left outside of the building and in these restrooms for participants to drop off their samples. If social distancing is required during this study, participants will be asked to collect the samples at home and drop them off in a cooler outside of the building to ensure social distancing. This subgroup will also complete additional 24-hour dietary recalls (study day 1, 42, 49, & 56).

Participants will continue to answer daily questionnaires until the third day of their third menstrual cycle, at which point they will discontinue answering questionnaires and consuming the study supplement. At the conclusion of the study, they will complete the final questionnaire that asks them which supplement they thought they were consuming to assess blinding efficacy. Participants will be instructed to return any unused supplements to the study site after the completion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Be a healthy female between the ages of 18 and 35 years who has regular menstrual cycles (i.e., every 24 to 33 days),
2. On the daily gastrointestinal symptom questionnaire for abdominal pain, participants must have a score of ≥ 3 for abdominal pain when thinking about their typical average score during first three days of menstruation,
3. Be on an combination oral contraceptive,
4. Willing and able to consume a probiotic or placebo supplement for approximately 8 weeks,
5. Willing and able to complete daily and weekly questionnaires online regarding dietary intake and general health and well-being, including gastrointestinal habits (Note: we will recruit participants who will have Internet access for the duration of the protocol, but understand that, once enrolled, situations may change. If this is the case, paper copies of the online forms will be provided.),
6. Willing to discontinue consumption of fermented foods or foods with live active cultures two weeks prior to beginning the study and throughout the study (This would include kefir, kombucha, yogurts with live, active cultures, etc.),
7. Willing to discontinue consumption of fiber supplements (This would include Metamucil, Benefiber, or other products with added fiber supplement.),
8. Willing to complete a pregnancy test before consuming the study supplement,
9. Willingness to complete questionnaires, records, and diaries associated with the study and to complete all study visits,
10. Able to provide informed consent,
11. Willing to provide a stool and vaginal sample ten times during the study (subgroup),
12. Typically have one stool per day (subgroup).

Exclusion Criteria:

1. Women who have a birth control implant, vaginal ring, shot, or patch or intrauterine device,
2. Women who are lactating, attempting to become pregnant, know that they are pregnant, or test positive on a pregnancy test,
3. Women who have consumed probiotic supplements in the last month,
4. Currently being treated for any physician-diagnosed diseases or conditions,
5. Women who have been diagnosed with any gynecological diseases of conditions (fibroma, endometriosis, etc),
6. Women who have pain that is caused by a disorder in the woman's reproductive organs. This would include a physician diagnosis such as endometriosis, adenomyosis, uterine fibroma, or a pelvic infection,
7. Allergy to milk, soy, or yeast,
8. Use of another investigational product within 3 months of the screening visit,
9. Use of any antibiotic drug within 1 month of screening.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participant must menstruate regularly and consume an oral contraceptive
Enrollment: 187 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Abdominal Pain | 28 days
  The primary outcome is the change (average of the first 3 days of the second menstrual cycle during the study when on the intervention minus the average of the first 3 days of the first menstrual cycle during the study prior to initiating the intervention) in the daily Visual Analog Score for abdominal pain between women on the probiotic versus the placebo interventions. The visual analog scale is scored between 0 (not pain at all) - 100 (worst pain imaginable). A higher score is less desirable. While we anticipate that a menstrual cycle should last 28 days, there may be variability in this number due to variability in the length of each participant's menstrual cycle.

SECONDARY OUTCOMES:
Menstrual Symptom Questionnaire | 28 days
  The Menstrual Symptom Questionnaire assesses symptoms related to each menstrual cycle.
Stool consistency | Each day up to 9 weeks
  Compare stool consistency, as measured by the Bristol Stool Form Scale (BSFS), between the probiotic and placebo groups. The BSFS is scored between 1 (hard stool) - 7 (liquid stool). A score of 4 or 5 is ideal.
Stool frequency | Each day up to 9 weeks
  Compare the number of stools between the probiotic and placebo groups.

OTHER OUTCOMES:
Digestive Health | Every 7 days up to 9 weeks
  Weekly GI symptoms assessed using the Gastrointestinal Symptom Rating Scale (GSRS). The GSRS consists of 15 questions related to 5 syndromes, constipation, diarrhea, reflux, abdominal pain, and indigestion. Symptoms are scored 1=no discomfort to 7=very severe discomfort. Scores from each of the 15 questions are summed for the total GSRS score.
Quality of Life Related to Digestive Health | Every 7 days up to 9 weeks
  Weekly GI experiences assessed using an in-house Digestion-Associated Quality of Life questionnaire.
Fecal microbial diversity | Every 7 days up to 9 weeks
  Changes in fecal microbial composition and diversity (i.e. alpha and beta diversity) will be assessed in a subgroup of participants.
Vaginal swab samples | Every 7 days up to 9 weeks
  Changes in vaginal microbial composition and diversity will be assessed in a subgroup of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Bobbi Langkamp-Henken, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Judkins TC, Oula ML, Sims SM, Langkamp-Henken B. The effect of a probiotic on gastrointestinal symptoms due to menstruation in healthy adult women on oral contraceptives: randomized, double-blind, placebo-controlled trial protocol. Trials. 2022 Jun 10;23(1):481. doi: 10.1186/s13063-022-06410-w. PMID 35689274